CLINICAL TRIAL: NCT00943527
Title: Molecular Breast Imaging: Effect of Menstrual Cycle, Hormone Therapy, and Tamoxifen on Tc-99m Sestamibi Uptake in the Breast.
Brief Title: Hormonal Effects on Tc-99m Sestamibi Uptake in the Breast
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Gamma Medica-Ideas (Industry)
Responsible Party: Principal Investigator, Deborah Rhodes, MD, Mayo Clinic
Other Study IDs: 07-004850
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Breast; Menstrual Cycle; Breast Cancer; Hormone; MBI; Molecular Breast Imaging; Breast Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Premenopausal Women who are not taking hormones or birth control. Ages 35-45 who have had a negative mammograph performed at the Mayo Clinic in Rochester within the last year.
- 2: Women Initiating Hormone Therapy and have had a negative mammogram preformed at the Mayo Clinic Rochester within the last year.
- 3: Women Initiating Tamoxifen who have had a negative mammogram preformed at the Mayo Clinic Rochester.

SUMMARY:
This study is to examine the effects of menstrual cycle, hormone therapy, and the use of tamoxifen on Tc-99m sestamibi uptake.

ELIGIBILITY:
Arm 1

Inclusion Criteria:

* age 35-45
* have regular menstrual cycles as defined by having menstrual cycle length of 25-31 days, with menstrual flow of 2-7 days, and no intermenstrual spotting or bleeding.
* have had a negative screening mammogram within one year prior to the MBI studies that is available for comparison.

Exclusion Criteria:

* currently using any exogenous hormones (e.g., hormonal contraceptives, sex steroid hormones) or any estrogen receptor modulating drugs (e.g., tamoxifen, raloxifene) or any aromatase inhibitors
* have a personal history of any cancer, except non-melanomatous skin cancer
* unable to understand and sign the consent form
* pregnant or lactating
* physically unable to sit upright and still for 30 minutes

Arm 2

Inclusion Criteria:

* scheduled to begin one of the following regimens of HT:
* Any dosage of any formulation of systemic estrogen therapy in the setting of a prior hysterectomy
* Any dosage of continuous estrogen plus monthly, cyclic progesterone therapy where the progesterone therapy is the oral, micronized formulation
* had a negative screening mammogram within one year prior to the MBI studies that is available for comparison.

Exclusion Criteria:

* have a personal history of any cancer, except non-melanomatous skin cancer
* unable to understand and sign the consent form
* pregnant or lactating
* physically unable to sit upright and still for 30 minutes

Arm 3

Inclusion Criteria:

* scheduled to begin treatment with tamoxifen Or are currently being treated with tamoxifen (for > 1 month) and have had an MBI scan performed prior to its initiation
* have had or will have the following test performed at Mayo Clinic: #87966, Cytochrome P450 2D6 genotyping for Tamoxifen Hormonal Therapy
* have had a screening or diagnostic mammogram within one year of the MBI studies that is available for comparison.

Exclusion Criteria:

* are using or have used any exogenous hormones (e.g., hormonal contraceptives, sex steroid hormones), any estrogen receptor modulating drugs other than tamoxifen, or any aromatase inhibitors from the time of 1 month prior to the first MBI until completion of the second MBI.
* have been treated or will be undergoing treatment with systemic chemotherapy or external radiation beam therapy to the breast from the time of 6 months prior to the first MBI until the completion of the second MBI.
* unable to understand and sign the consent form
* pregnant or lactating
* physically unable to sit upright and still for 30 minutes

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States